CLINICAL TRIAL: NCT00497926
Title: Induction of Donor Specific Tolerance in Recipients of Living Kidney Allografts by Donor FCRx Infusion
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: living donor kidney program terminated due to slow pace of phase 3 study enrollment
Sponsor: Talaris Therapeutics Inc. (Industry)
Collaborators: Northwestern University (Other); Regenerex, LLC (Unknown); Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FCR001A2201
Record Dates: First submitted 2007-07-06; First posted 2007-07-09 (Estimated); Last update posted 2023-10-11 (Actual); Status verified 2023-10

CONDITIONS: Kidney Failure
Keywords: Kidney transplant; Tolerance; Marrow/Enriched Hematopoietic Stem Cell Transplant
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Living Kidney Allograft (Experimental): Recipients with the need for a living kidney allograft are treated with an enriched hematopoietic stem cell infusion from the same living donor
  Interventions: Biological: Enriched Hematopoietic Stem Cell Infusion

INTERVENTIONS:
Biological: Enriched Hematopoietic Stem Cell Infusion — Enriched Hematopoietic Stem Cell Infusion

SUMMARY:
An open-label study to assess the safety, efficacy, and tolerance of FCRx cell therapy in adult recipients within 12 months after kidney transplantation from a living donor.

DETAILED DESCRIPTION:
Research study which involves the use of a combination of an Enriched Hematopoietic Stem Cell Infusion (stem cells, produced by the bone marrow, generate the cells that form the blood elements, help fight infection and assist in clotting) and kidney transplantation from the same donor to try to avoid the need for long-term anti-rejection drug therapy. The desired result of this study is to allow the body to develop "tolerance" to the transplanted kidney. Tolerance means that the body would see the transplanted kidney as part of the patient and not try to get rid of, or reject it. To prevent rejection, drugs called immunosuppressive agents must be taken on a daily basis. The purpose of this study is to determine if this procedure is safe and to try to substantially reduce or even eliminate the need for anti-rejection medications.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be between the ages of 18 and 65 years and meet the institution's criteria for renal transplantation for end-organ failure
* Meets the transplant criteria by the study site and both the recipient and donor have been accepted as candidates for standard of care living kidney donation and transplantation
* Patient is receiving a renal transplant only
* The crossmatch is negative between donor and recipient. An initial crossmatch will be performed prior to stem cell mobilization to determine if subject can proceed with the apheresis.
* Potential recipients who are women of child bearing potential must have a negative pregnancy test (urine test is acceptable) within 48 hours prior to receiving Granulocyte colony-stimulating factor (G-CSF) and agree to use reliable contraception for 1 year following FCRx infusion
* Potential donors who are women of child bearing potential must have a negative pregnancy test (urine test is acceptable) within 48 hours prior to receiving G-CSF
* No evidence of donor-specific antibody presently or historically
* Panel Reactive Antibody (PRA) less than or equal to 20

Note: The subjects do not need to be local residents in order to be eligible for this trial, but must be willing to reside in the area, or within a four-hour drive, for the first month of the protocol so that they can be monitored closely in the early post-transplant period.

Exclusion Criteria:

* Clinically active bacterial, fungal, viral or parasitic infection
* Pregnancy
* Clinical or serologic evidence of viral infection which would preclude the recipient from receiving a kidney transplant or FCRx infusion
* Previous radiation therapy at a dose which would preclude Total Body Irradiation (TBI)
* Positive crossmatch between donor and recipient
* Evidence for immunologic memory against donor
* Body Mass Index (BMI) >35 or <18
* Positive serologies for Hepatitis B Virus (HBV), Hepatitis C Virus (HCV), human immunodeficiency virus (HIV)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2008-03 (Actual); Primary Completion 2023-03 (Actual); Study Completion 2023-04 (Actual)

PRIMARY OUTCOMES:
Enriched Hematopoietic Stem Cell Engraftment | One month to three years

CONTACTS AND LOCATIONS:
Overall Officials: Ken Abrams, MD, Study Director — Talaris Therapeutics
Locations (2):
- United States (2):
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Duke University, Durham, North Carolina

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Leventhal JR, Galvin J, Ison MG, Feng CY, Ding R, Lee JR, Li C, Mathew JM, Gallon L, Gibson M, Belshe D, Tollerud DJ, Gornstein E, Suthanthiran M, Ildstad ST. Evaluation of Immunocompetence and Biomarkers of Tolerance in Chimeric and Immunosuppression-free Kidney Allograft Recipients. Transplantation. 2023 Oct 1;107(10):e257-e268. doi: 10.1097/TP.0000000000004666. Epub 2023 Sep 25. PMID 37370204
- [Derived] Gallon L, Mathew JM, Bontha SV, Dumur CI, Dalal P, Nadimpalli L, Maluf DG, Shetty AA, Ildstad ST, Leventhal JR, Mas VR. Intragraft Molecular Pathways Associated with Tolerance Induction in Renal Transplantation. J Am Soc Nephrol. 2018 Feb;29(2):423-433. doi: 10.1681/ASN.2017030348. Epub 2017 Nov 30. PMID 29191961
- [Derived] Leventhal JR, Elliott MJ, Yolcu ES, Bozulic LD, Tollerud DJ, Mathew JM, Konieczna I, Ison MG, Galvin J, Mehta J, Badder MD, Abecassis MM, Miller J, Gallon L, Ildstad ST. Immune reconstitution/immunocompetence in recipients of kidney plus hematopoietic stem/facilitating cell transplants. Transplantation. 2015 Feb;99(2):288-98. doi: 10.1097/TP.0000000000000605. PMID 25594553